CLINICAL TRIAL: NCT03434197
Title: Randomized Controlled Study to Evaluate the Safety and Efficacy of SFPP in Knee Osteoarthritis Using Diclofenac Gel as the Comparator
Brief Title: Safety and Efficacy of SFPP in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPJ.01.2017
Record Dates: First submitted 2018-02-02; First posted 2018-02-15 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis Knee Pain
Keywords: Osteoarthritis Knee Pain
MeSH Terms: interventions — diclofenac diethylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFPP (Esflurbiprofen plaster) (Experimental): A plaster containing 40 mg of Esflurbiprofen and 36.2 mg of Japanese Pharmacopoeia mentha oil per patch (10 × 14 cm)
  Interventions: Drug: Esflurbiprofen
- Diclofenac gel (Active Comparator): A gel containing 11.6 mg of Diclofenac diethylamine (equivalent to 10 mg of diclofenac sodium) per 1 g (1 tube contains 20 g)
  Interventions: Drug: Diclofenac diethylamine

INTERVENTIONS:
Drug: Esflurbiprofen — A plaster containing 40 mg of Esflurbiprofen and 36.2 mg of Japanese Pharmacopoeia mentha oil per patch (10 × 14 cm)
  Arms: SFPP (Esflurbiprofen plaster)
Drug: Diclofenac diethylamine — A gel containing 11.6 mg of Diclofenac diethylamine (equivalent to 10 mg of diclofenac sodium) per 1 g (1 tube contains 20 g)
  Arms: Diclofenac gel

SUMMARY:
The objectives of this study are to demonstrate the non-inferiority of esflurbiprofen plaster (SFPP) 40 mg applied for 2 weeks to diclofenac gel, the comparator, in terms of efficacy in patients with knee osteoarthritis (OA) and to examine the safety of SFPP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had unilateral knee pain and were classified as Grade II or III according to Kellgren-Lawrence (KL) grading and whose non-assessed knee is not graded higher than the assessed knee based on x-ray in standing, weight-bearing extension position within 90 days before screening visit (1st visit)
* Patients whose knee pain on rising from the chair assessed by visual analogue scale (rVAS) of the assessed knee meets all the following criteria for the level of pain; < 80 mm at washout visit (2nd visit), ≥ 40 mm at baseline visit (3rd visit), Worsening of ≥ 15 mm at baseline visit (3rd visit) compared with rVAS at washout visit (2nd visit) as a result of discontinuation of use of NSAIDs

Exclusion Criteria:

* Patients with complication of rheumatoid arthritis, history of knee surgery, malignant tumor, neuropsychiatric disease, or serious disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Improvement of Knee pain on rising from the chair | 5 weeks (3 weeks of observation period and follow up with 2 weeks treatment period)
  0-100 mm Visual Analogue Scale (VAS) (0mm, no pain; 100mm, worst pain ever)

SECONDARY OUTCOMES:
Improvement of Changes in total clinical symptom | 5 weeks (3 weeks of observation period and follow up with 2 weeks treatment period)
  Assessment from investigator ( 0=Absent, 1=Mild, 2=Moderate, 3=Severe; total= 0 - 45 )
Improvement of Investigator's global assessment | Last visit
  Investigator's global assessment Questionnaire ( 1=Marked, 2=Moderate, 3=Mild, 4=No change, 5=Worse)
Improvement of Patient's global assessment | Last visit
  Patient's global assessment Questionnaire ( 1=Marked, 2=Moderate, 3=Mild, 4=No change, 5=Worse )
Improvement of Knee pain on walking | 5 weeks (3 weeks of observation period and follow up with 2 weeks treatment period)
  0-100 mm Visual Analogue Scale (VAS) (0mm, no pain; 100mm, worst pain ever)
Number of Rescue drug use during treatment period | 3 weeks (1 weeks of observation period and follow up with 2 weeks treatment period)
  Report from investigator
Number of Adverse events and adverse drug reactions | 5 weeks (3 weeks of observation period and follow up with 2 weeks treatment period)
  Report from investigator

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Setyohadi, Dr. Sp.PD-KR, Study Chair — Rumah Sakit Cipto Mangunkusumo; Sumariyono, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit Cipto Mangunkusumo; Tanggo Meriza, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit Islam Pd. Kopi; Sandra Sinthya Langow, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit Siloam Karawaci; Ika Wulan Yuliani, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit Anna Medika Bekasi; Sumartini Dewi, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit Hasan Sadikin; Andri Reza, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit Umum Daerah Al Ihsan Bale Endah; Laniyati Hamijoyo, Dr. Sp.PD-KR, Principal Investigator — Klinik Perisai Husada; Yuliasih, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit UD Dr. Soetomo; Lita Diah Rahmawati, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit TNI AU Soemitro; Cesarius Singgih Wahono, Dr. Sp.PD-KR, Principal Investigator — Rumah Sakit UD Dr. Saiful Anwar; Handono Kalim, Dr. Sp.PD-KR, Principal Investigator — Rheumatology and Allergy Clinic
Locations (11):
- Indonesia (11):
  - Klinik Perisai Husada, Bandung
  - Rumah Sakit Hasan Sadikin, Bandung
  - Rumah Sakit Umum Daerah Al Ihsan Bale Endah, Bandung
  - Rumah Sakit Anna Medika Bekasi, Jakarta
  - Rumah Sakit Cipto Mangunkusumo, Jakarta
  - Rumah Sakit Islam Pd. Kopi, Jakarta
  - Rumah Sakit Siloam Karawaci, Jakarta
  - Rheumatology and Allergy Clinic, Malang
  - Rumah Sakit UD Dr. Saiful Anwar, Malang
  - Rumah Sakit TNI AU Soemitro, Surabaya
  - Rumah Sakit UD Dr. Soetomo, Surabaya

IPD SHARING:
Plan to Share IPD: No